CLINICAL TRIAL: NCT06100445
Title: Barriers and Facilitators to Exercise Engagement in People Over 60 at Risk of Falls: an Exploratory Study
Brief Title: Exercise Engagement in People Over 60 at Risk of Falls
Status: Recruiting | Type: Observational
Sponsor: East Lancashire Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Michelle Thirlwall, Principal Investigator, East Lancashire Hospitals NHS Trust
Other Study IDs: DEV072
Record Dates: First submitted 2023-10-13; First posted 2023-10-25 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Musculoskeletal Injury; Frailty; Physical Inactivity; Health Behavior
MeSH Terms: conditions — Frailty; Sedentary Behavior; Health Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Semi structured interviews — Gaining qualitative data

SUMMARY:
It is a qualitative study, using semi structured interviews to explore patient's experiences of falls and their perceptions on facilitators and barriers to exercise.

Aim: To explore reasons for and against engaging with exercises at home in participants over the age of 60 at risk of falls.

To explore:

1. Patients' preferences to exercise format and type eg/ leaflet, online, access, such as the Chartered Society of Physiotherapy (CSP) chair exercises leaflet or individual personalized rehabilitation programme handouts
2. The ability to discuss falls risk with health professionals.
3. If health inequalities exist with people at risk of falls and exercising.
4. Sustainability of exercise, in order to reduce the risk of falls in this population.
5. The need to develop MSK internal and external facing falls management pathways.

Suitability: Patients over the age of 60, who have been identified at risk of falls, having been referred to MSK Physiotherapy in Rossendale.

'Risk of falls' is defined as: patient self-reports they are unsteady, had one or more fall in the last 6 months, or clinician identified a slow/unsteady gait pattern on examination.

Semi structured interviews on up to ten participants. It is anticipated that this sample size will give adequate data saturation. Approximately 12 months from participant recruitment to analysis of findings.

DETAILED DESCRIPTION:
One in three people over the age of 65 and one in two over the age of 80 will fall each year. A fall is the main reason older people attend A and E. Falls can result in soft tissue injuries and broken bones, the most significant being a hip fracture, and these often require physiotherapy input. Locally, we have above average rates of hip fracture. Falling also reduces confidence and further mobility, which can also impact on developing long term health conditions.

Research has shown that exercise can help improve the strength and balance in people over 60 at risk of falls. Balance and strength exercises have been shown in previous research to reduce the risk of falls by 25% in patient's over 60. However, in other research, 78% of patients over the age of 75 have not done exercises at home in the last 5 years.

Exploring patient views on exercises and their physiotherapy experience will help us understand why patients engage or not with exercise and improve our services.

Patients who are at risk (identified through the EMIS template) of falls and have expressed an interest in being involved in research and who meet the additional eligibility criteria will be approached by the researcher. Eligible participants interested in participating will be contacted and sent the patient information sheet and consent form. They will be contacted within two weeks to see if they want to participate and assistance with the consent form either over phone or face to face.

A copy of the consent form will be scanned into the participant notes on EMIS, and paper copies stored securely in a locked filing cabinet.

All participants will have the opportunity to ask any questions regarding consent and the study prior to commencing the interviews and data collection.

The right of the participant to refuse to participate in research study without giving reasons will be respected. All participants are free to withdraw at any time without giving reasons and without prejudicing further treatment.

Face to face interviews will be recorded via an encrypted voice Dictaphone recorder. If conducting interviews via telephone call or MS teams, then voice recordings using the encrypted dictaphone will also be used. The interview will take approximately half an hour, and patients will only be interviewed once, there will be no follow up in this study.

All participant identifiable information will be kept confidential, and a participant number will be used. Recordings will be loaded onto a password protected secure trust server, accessible only to the researcher and the original recording deleted off the Dictaphone within 48 hours (about 2 days). Once transcribed, the recording on the drive will then be deleted.

Anonymised qualitative data will be transcribed by an NIHR transcriber. Then it will be analysed using thematic analysis using NVivo version 12, or the most up to date version of NVivo, a qualitative data analysis software. All data will be anonymised prior to analysis using an allocated participant ID number.

In the unlikely event that distress will be identified, the interview will be stopped, and the reason for the distress dealt with as per normal clinical practice. The participant will be given the option to stop participating (see withdrawal from participating below), or to continue with the interview at a later time. Participants can withdraw at any time up to once the interviews have been transcribed.

Data will then be used to improve patient services in physiotherapy, as well as highlight any service pathway and health inequality needs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or over
* At risk of falls or had a fall due to a musculoskeletal cause (pain, muscle weakness, balance issue)
* Has capacity to consent, as deemed by the direct care team and researcher
* Can communicate in English OR the use of a translation service - Able to independently participate in an interview either face-to-face or via remote means OR can use a translation service

Exclusion Criteria:

- Aged under 60

* Have a medical cause of falls OR currently under investigation for a medical cause of falls (eg/ dizziness, cardiac, visual impairment reported as being the cause of the fall as opposed to weakness or pain in lower limbs/balance issues or unsteady on feet)
* Moderate to severe cognitive impairment impairing capacity to consent

Ages: 60 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a single centre study, based at Rossendale Health Centre. The MSK Physiotherapy Service is part of an integrated model in East Lancashire Hospitals NHS Trust (ELHT) for managing musculoskeletal, rheumatology, orthopaedic and pain conditions (https://elht.nhs.uk/services/integrated-msk-pain-and-rheumatology-service). The aim is to deliver the highest quality of care and support for patients with musculoskeletal conditions. This includes patients who have been referred following falls resulting in fractures or soft tissue injuries, and painful long-term conditions such as osteoarthritis which can impact mobility. A third of the caseload in MSK physiotherapy consists of patients over the age of 60.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Explore reasons for and against engaging with exercises at home. | Through study completion, an average of 1 year
  By identifying themes during anaylsis of study interviews

SECONDARY OUTCOMES:
Patients' thoughts on service materials, provision and communication | Through study completion, an average of 1 year
  Identify preferred exercise format and understanding of information eg/ leaflet, online, access, such as the Chartered Society of Physiotherapy (CSP) chair exercises leaflet or their own online personalised rehabilitation programme handouts by analysing themes of the interviews

CONTACTS AND LOCATIONS:
Overall Officials: James Boateng, Study Chair — East Lancashire Hospitals NHS Trust; Elizabeth Lightbody, Study Chair — National Institute for Health Research, United Kingdom
Locations (1):
- East Lancashire Hospitals NHS Trust, Blackburn, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Older adult perceptions of exercise in the community — https://research.monash.edu/en/publications/older-adult-perceptions-of-participation-in-group-and-home-based-
- See also: National falls data and fragility priority and frameworks — https://www.gov.uk/government/publications/falls-applying-all-our-health/falls-applying-all-our-health
- See also: NICE guidelines, updated 2024 — https://www.nice.org.uk/guidance/cg161
- See also: WHO guidelines — https://www.who.int/teams/social-determinants-of-health/safety-and-mobility/step-safely